CLINICAL TRIAL: NCT01665300
Title: Usefulness of Myocardial Deformation Imaging in Breast Cancer Patients Treated With Trastuzumab for Early Detection of Myocardial Dysfunction
Brief Title: Usefulness of Myocardial Deformation Imaging for Trastuzumab-induced Cardiotoxicity
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Kwan Kim, MD, PhD, Assistant Professor, Seoul National University Cardiovascular center, Seoul National University Hospital
Other Study IDs: H1106-026-365
Record Dates: First submitted 2011-12-13; First posted 2012-08-15 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Left Ventricular Function Systolic Dysfunction; Cardiotoxicity
Keywords: myocardial deformation imaging; Trastuzumab
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — genetic susceptibility for HER2(+)cardiotoxicity
Oversight: Data Monitoring Committee: No

SUMMARY:
Trastuzumab prolongs survival in patients with human epidermal growth factor receptor type 2-positive breast cancer. Sequential left ventricular (LV) ejection fraction (EF) assessment has been mandated to detect myocardial dysfunction because of the risk of heart failure with this treatment. Myocardial deformation imaging is a sensitive means of detecting LV dysfunction, but this technique has not been evaluated in patients treated with trastuzumab. The aim of this study was to investigate whether changes in tissue deformation, assessed by myocardial strain and strain rate (SR), are able to identify LV dysfunction earlier than conventional echocardiographic measures in patients treated with trastuzumab.

DETAILED DESCRIPTION:
The investigators will prospectively evaluate whether changes in tissue deformation, assessed by myocardial strain and strain rate (SR) and identify possibility of early detection of LV dysfunction in patients treated with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* HER2(+) breast cancer, anticipating Trastuzumab therapy

Exclusion Criteria:

* Refusal to informed consent
* Congenital heart disease
* Significant arrhythmia in EKG
* Regional wall motion abnormality (+) in echocardiography
* Poor sonic window

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators evaluated serial echocardiograms (baseline, 3, 6, 9, and 12 months)from 120 consecutive female patients receiving trastuzumab as part of their treatment for either early or advanced breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
LV systolic dysfunction | 3-month F/U
  LV systolic dysfunction was defined as following;
  1. An EF unit drop of ≥10% from the baseline available echocardiogram or
  2. Change in strain or strain rate : drop(decrement) corresponding to ≥1 SD of the relevant parameter assessed at the baseline available echocardiogram

SECONDARY OUTCOMES:
LV systolic dysfunction | 6,9, and 12-month F/U
  LV systolic dysfunction was defined as following;
  1. An EF unit drop of ≥10% from the baseline available echocardiogram or
  2. Change in strain or strain rate : drop(decrement) corresponding to ≥1 SD of the relevant parameter assessed at the baseline available echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Kwan Kim, M.D., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea